CLINICAL TRIAL: NCT01093300
Title: Comparison of the Efficacy of Paclitaxel-releasing Balloon Catheter System Versus the Everolimus-Eluting Stent System for Treatment of In-Stent Restenosis Lesions - Harmonizing Optimal Strategy for Treatment of In-Stent Restenosis Lesions (The HOST-ISR Trial) -
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Seoul National University Hospital IRB, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HOST-ISR trial
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Last update posted 2023-04-20 (Actual); Status verified 2013-03

CONDITIONS: In-stent Restenosis Lesion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel-eluting balloon catheter (Experimental): Paclitaxel-eluting balloon catheter use for treatment of ISR lesion
  Interventions: Device: Paclitaxel-eluting balloon catheter
- Everolimus-eluting stent (Active Comparator): Everolimus-eluting stent use for treatment of ISR lesion
  Interventions: Device: Everolimus-eluting stent

INTERVENTIONS:
Device: Paclitaxel-eluting balloon catheter
  Arms: Paclitaxel-eluting balloon catheter
Device: Everolimus-eluting stent
  Arms: Everolimus-eluting stent

SUMMARY:
In-stent restenosis (ISR) lesions are considered one of the toughest lesions that interventional cardiologists encounter in the drug eluting stent (DES) era. The current consensus in treating ISR is implantation of another DES into the restenosed segment. However the recent results of paclitaxel-releasing balloon catheter (PRBC) in ISR lesions have been very encouraging. The aim of HOST-ISR trial is to investigate the efficacy and safety of PRBC compared with everolimus-eluting stent (EES) in preventing neointimal growth in ISR lesions. HOST-ISR trial is a multicenter, open-label, prospective, randomized trial to test whether PRBC is non-inferior to EES in preventing neointimal growth in ISR lesions. It plans to enroll a total of 264 patients with ISR, randomizing the cohort 1:1 to either PRBC or EES. The primary endpoint will be in-segment late luminal loss at 9 months angiographical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18y
* Significant ISR lesion (>50% by visual estimate) of previously stented de novo coronary artery
* Evidence of myocardial ischemia (e.g., stable, unstable angina, recent infarction, silent ischemia, positive functional study or a reversible changes in the electrocardiogram (ECG) consistent with ischemia) or ISR with diameter stenosis > 70%
* Written, informed consent
* Target lesion(s) located in a native coronary artery within a previously stented lesion with previous stent diameter of ≥ 2.5 mm and ≤ 4.00 mm
* Target lesion(s) amenable for percutaneous coronary intervention

Exclusion Criteria:

* Hypersensitivity to aspirin, clopidogrel, heparin, sirolimus, paclitaxel or radiocontrast media
* Systemic sirolimus use within 12 months
* Female of childbearing potential
* History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia)
* Gastrointestinal or genitourinary bleeding within the prior 3 months, or major surgery within 2 months
* Non-cardiac co-morbid conditions present with life expectancy <1 year or that may result in protocol non-compliance
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period
* ISR of left main coronary artery
* Restenosis of two stented bifurcation lesion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)

PRIMARY OUTCOMES:
Late luminal loss in the analysis segment | 9 months
  Analysis segment is defined as +/- 5mm of the previous stented/inflated segment of the vessel

SECONDARY OUTCOMES:
Late luminal loss in the inflation/in-stent segment | 9 months
Target lesion/vessel revascularization, myocardial infarction | 1, 2 years
Periprocedural myocardial infarction | 3 days
% diameter stenosis in the analysis segment & in the inflation/in-stent segment | 9 months
Neointimal volume, % neointimal volume, % volume obstruction | 9 months
  The above parameters will be assessed by IVUS
Time interval from device insertion to initiation of deployment | 0 days
Stent thrombosis | 1, 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea